CLINICAL TRIAL: NCT05139433
Title: Brief Internet-delivered Cognitive-behavioral Intervention for Children and Adolescents With Anxiety and Depression Symptoms During the COVID-19 Pandemic: a Randomized Clinical Trial
Brief Title: Brief Internet-delivered Intervention for Children and Adolescents With Anxiety and Depression Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Guilherme Vanoni Polanczyk, MD PhD, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Proc. FAPESP 2016/22455-8
Record Dates: First submitted 2021-11-04; First posted 2021-12-01 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Childhood Anxiety Disorder; Childhood Depression
Keywords: Children; Anxiety; Depression; Stress; Cognitive Behavioral Therapy; Telemedicine; Irritability; Covid-19 pandemic; Adolescents
MeSH Terms: conditions — Anxiety Disorders; Depression; COVID-19 | interventions — Mental Health Teletherapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to be either in the intervention group (internet-based therapy) or the active control group (educational videos)
Who Masked: Outcomes Assessor
Masking Description: A trained clinical psychologist, blinded to which group the subject was allocated, will clinically assess the child/adolescent at T0, T1 and T2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this arm will receive 5 internet-delivered cognitive-behavioral intervention and will have access to 15 educational videos
  Interventions: Behavioral: Telepsychotherapy; Behavioral: Psychoeducational Videos
- Active Control Group (Active Comparator): Participants in this arm will have access to 15 educational videos.
  Interventions: Behavioral: Psychoeducational Videos

INTERVENTIONS:
Behavioral: Telepsychotherapy — 5 weekly psychotherapy sessions that will cover the following contents: psychoeducation on stress responses, family communication, relaxation and mindful techniques, emotion recognition, management of irritability, behavioral activation and cognitive restructuring. The sessions will be implemented via the internet by a trained psychologist. Participants will also have access to the psychoeducational videos described at "intervention 2"
  Arms: Intervention Group
Behavioral: Psychoeducational Videos — 15 educational videos to be watched by the families. There will be one video about psychoeducation on stress responses, one about family communication, four about mindfulness and relaxation techniques, two about emotion recognition, one about management of irritability, one about behavioral activation, three about healthy routines, one about cognitive restructuring, and one about management of anxiety crisis.

SUMMARY:
Investigators developed a brief standardized internet-delivered cognitive-behavioral program for treating anxious and depressive symptoms in children and adolescents in the context of COVID-19 pandemics in Brazil. A 2-arm parallel-randomized controlled clinical trial will be conducted to test the efficacy of this program (intervention group), in comparison with a educational-only intervention program based on videos (active control group). 280 children and adolescents (8 to 17 years-old) with clinically significant anxious and/or depressive symptoms will be recruited through internet and social media. They will be randomized either to the intervention (n=140) or active control group (n=140). Participants will be recruited from across the country. The therapeutic program consists of 5 weekly sessions covering the following contents: education on stress reactions, family communication, relaxation and mindful techniques, emotion recognition, management of irritability, behavioral activation, and cognitive restructuring. The educational program consists of 15 videos covering the same content. Participants in the intervention group will also have access to these videos. Both child/adolescent and at least one caregiver will be required to take part in the sessions (and watch the videos). Participants will be assessed at the beginning (baseline; T0) at the end (endpoint; T1), and 30 days after the intervention (follow-up; T2) with standardized questionnaires, through an interview with a blinded investigator. Participants that develop severe symptomatology requiring further support during the intervention (such as psychiatric pharmacological treatment and/or more intensive psychotherapy) will be referred to adequate treatment. During the week prior to the intervention and the first week after its end, adolescents (older than 12 years-old) in both groups with access to a smartphone will be asked to report their momentary mood, emotions, and stress several times a day using the same smartphone app that will deliver the educational content to both groups. Adolescents will also be asked to install a second smartphone application that captures data from the phone sensors to provide proxies on behaviors associated with depression, such as social isolation (by the proximity with other devices, time spent on social media, as well as environmental sound and light) amount of inactivity (by assessing the maximum distance traveled throughout the day), among others.

DETAILED DESCRIPTION:
Investigators developed a brief standardized and manualized internet-delivered cognitive-behavioral (iCBT) program for treating anxious and depressive symptoms in children and adolescents in the context of COVID-19 pandemics in Brazil, to be implemented by trained psychologists. A 2-arm parallel-randomized controlled clinical trial (RCT) will be conducted to test the efficacy of this program (intervention group), in comparison with a educational-only intervention program based on videos (active control group). 280 children and adolescents (8 to 17 years-old) with clinically significant anxious and/or depressive symptoms (total t-score of 70 or above in the parent and child report versions of the 25-item Revised Children's Anxiety and Depression Scale) will be recruited through internet and social media. They will be randomized either to the intervention (n=140) or active control group (n=140). Since all interventions will be conducted online, participants will be recruited from across the country. The therapeutic program consists of 5 weekly sessions delivered to children or adolescents and their parents and covering the following contents: education on stress reactions, family communication, relaxation and mindful techniques, emotion recognition, management of irritability, behavioral activation, and cognitive restructuring. All sessions will be recorded and 10% of them will be randomly selected to be watched by one of the authors of the psychotherapeutic program to assess protocol adherence. The educational program consists of 15 videos covering the same content. Participants in the intervention group will also have access to these videos. Both child/adolescent and at least one caregiver will be required to take part in the sessions (and watch the videos). Participants in both groups will be assessed at the beginning (baseline; T0) at the end (endpoint; T1), and 30 days after the intervention (follow-up; T2) with standardized questionnaires, through an interview with a blinded investigator at T0, T1, and T2. Participants that develop severe symptomatology requiring further support during the intervention (such as psychiatric pharmacological treatment and/or more intensive psychotherapy) will be referred to adequate treatment. During the week prior to the intervention and the first week after its end, adolescents (older than 12 years-old) in both groups who have access to a smartphone will be asked to report their momentary mood, emotions, and stress several times a day using the same smartphone app that will deliver the educational content to both groups. Adolescents will also be asked to install a second smartphone application that captures data from the phone sensors to provide proxies on behaviors associated with depression, such as social isolation (by the proximity with other devices, time spent on social media, as well as environmental sound and light) amount of inactivity (by assessing the maximum distance traveled throughout the day), among others.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged between 8-17 years;
* Living in Brazil
* Total t-score of 70 or above in the 25-item version of the Revised Children's Anxiety and Depression Scale - parent report and child report versions

Exclusion Criteria:

* No contact between child/adolescent and parents in the 15 days previous to the beginning of the intervention
* Unavailability of at least one parent/caregiver to participate in all of the telepsychotherapeutic sessions (intervention group) or watch the videos along their child (active control group)
* Inability of the caregivers to understand the parent-report scales or the content of the interventions, according to the clinical judgement of a clinical psychologist
* Indications that the child might have a severe mental disorder and/or social condition that require a more intensive assessment and treatment, such as autism spectrum disorder, severe mood disorder, suicide risk, schizophrenia, intellectual disability, intense intrafamiliar conflict or intense maltreatment victimization, according to the clinical judgement of a clinical psychologist; suicidality will be assessed with the aid of the 4 questions of the Mood and Feelings Questionnaire (MFQ) questionnaire that focus on this trait ("S/he thought that life wasn't worth living", "S/he thought about death or dying", "S/he thought his/her family would be better off without him/her", "S/he thought about killing him/herself") (individuals that answer "yes" to the last question will be excluded from the study and referred to adequate and more intensive care)
* Current use or in the last 1 month of any psychiatric medication or psychotherapy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Anxiety and depressive symptoms at T1- caregiver report | At entry (T0), 1-3 days after the last psychotherapeutic session (intervention group) OR 1-3 days after the last video is made available (active control group)
  The first primary outcome is the change in depressive and anxiety symptomatology, measured by the 25-item version of the Revised Children's Anxiety and Depression Scale, parent reported, between T0 and T1. The RCADS is a 25-item scale that measures the frequency of anxiety and low mood symptoms using a 4-point Likert scale ("never", "sometimes", "often", and "always") based on personal observations from parents or legal guardians. The scale has two subscales assessing Anxiety and Depression, and an overall score. It will be completed by an independent clinician blinded to allocation based on an interview with the main caregiver (through videoconference or phone call).
Anxiety and depressive symptoms at T1 - child/adolescent report | At entry (T0), 1-3 days after the last psychotherapeutic session (intervention group) OR 1-3 days after the last video is made available (active control group)
  The change in depressive and anxiety symptomatology, measured by the 25-item version of the Revised Children's Anxiety and Depression Scale (RCADS), child reported, between T0 and T1. This version of RCADS is a 25-item scale that measures the frequency of anxiety and low mood symptoms using a 4-point Likert scale ("never", "sometimes", "often", and "always") based on personal observations from the child. The scale has two subscales assessing Anxiety and Depression, and an overall score.It will be completed by an independent clinician blinded to allocation based on an interview with the child/adolescent (through videoconference or phone call).

SECONDARY OUTCOMES:
anxiety and depressive symptoms at T2 - parent report | At entry (T0) and 30 days after the last psychotherapeutic session (intervention group) or 30 days after the last video is made available (active control group) (T2)
  The first secondary outcome is the change in depressive and anxiety symptomatology, measured by the 25-item version of the Revised Children's Anxiety and Depression Scale, parent report, between T0 and T2. This version of RCADS is a 25-item scale that measures the frequency of anxiety and low mood symptoms using a 4-point Likert scale ("never", "sometimes", "often", and "always") based on personal observations from parents or legal guardians. The scale has two subscales assessing Anxiety and Depression, and an overall score.
  It will be fulfilled by the blind assessor, in an interview with the main caregiver (through videoconference or phone call).
anxiety and depressive symptoms at T2 -- child/adolescent report | At entry (T0) and 30 days after the last psychotherapeutic session (intervention group) or 30 days after the last video is made available (active control group) (T2)
  The change in depressive and anxiety symptomatology, measured by the 25-item version of the Revised Children's Anxiety and Depression Scale (RCADS), child reported, between T0 and T2. This version of RCADS is a 25-item scale that measures the frequency of anxiety and low mood symptoms using a 4-point Likert scale ("never", "sometimes", "often", and "always") based on personal observations from the child. The scale has two subscales assessing Anxiety and Depression, and an overall score. It will be completed by an independent clinician blinded to allocation based on an interview with the child/adolescent (through videoconference or phone call).
The Clinical Global Impressions Scale | At entry (T0), 1-3 days after the last psychotherapeutic session (intervention group) OR 1-3 days after the last video is made available (active control group) (T1) and 30 days after these dates (T2)
  The blind assessor will evaluate the global functioning of the child/adolescent by an interview with the main caregiver and the child/adolescent (through videoconference or phone call) assessing the difference in scoring of the Clinical Global Impressions Scale - Severity (CGI-S) between T0 and T1 and T0 and T2 and the scoring of the Clinical Global Impressions Scale - Improvement (CGI-I) at T1 and T2. Scores of CGIS range from 1 to 7 (with higher scores corresponding to more intense symptomatology). Scores of CGI-I also range from 1 ("very much improved") to 7 ("very-much worse")
Children's Global Assessment Scale (CGAS) | At entry (T0), 1-3 days after the last psychotherapeutic session (intervention group) OR 1-3 days after the last video is made available (active control group) (T1) and 30 days after these dates (T2)
  the blind assessor will evaluate the global functioning of the child/adolescent by an interview with the main caregiver and the child/adolescent (through videoconference or phone call) assessing the difference in the scores of the Children's Global Assessment Scale (CGAS) at T0 and T1, and T0 and T2. CGAS scoring ranges from 0 to 100, with higher scores indicating better functionality.
impact of mental health symptomatology | At entry (T0), 1-3 days after the last psychotherapeutic session (intervention group) OR 1-3 days after the last video is made available (active control group) (T1) and 30 days after these dates (T2)
  The change of the impact of the child/adolescent mental health symptomatology between T0 and T1, and T0 and T2 will be assessed using the Strengths and Difficulties Questionnaire (SDQ) Impact Scale. Its score ranges from 0 to 10, with higher scores indicating greater severity of distress and impairment. It will be fulfilled by the blind assessor, in an interview with the main caregiver and the child/adolescent (through videoconference or phone call).
Ecological Momentary Assessment of Emotional Problems | During the week prior to the beginning of the intervention and during the week after it
  Adolescents (12years-old or older) in both groups with access to a smartphone will complete a brief, in-the-moment assessment of emotions, mood, stress, and anxiety. Participants will receive a notification in their smartphone to answer a series of questions intended to reflect their current state ("Right now, I feel…"), with a 7-point Likert scale answer options (0 = Not at all, 7 = Very much). This Experience Sampling Method (ESM) schedule consists of 17 questions, taking up to 3min to complete. The ESM schedule will be delivered four random times per day within four three-hour blocks from 9:00 to 21:00 for six consecutive days in the week prior to the beginning of the intervention (first session, in the Intervention Group, and the availability of the first video, in the Active Control Group) and the week after the end of it (therefore, pre and post intervention).
Passive data collection | During the 5 weeks of the intervention until 30 days after the last psychotherapeutic session (intervention group) or 30 days after the last video is made available (active control group)
  Adolescents (12years-old (or older) in both groups with access to a smartphone will be asked to install the pRMT app from RADAR-base. This app will run in the background, requiring minimal input from participants and will use the phone sensors to collect data on: a) ambient noise and light; b) relative GPS location (that is, the amount of distance travelled, not absolute coordinates or precise geographical location); c) bluetooth connectivity; d) length and duration of calls; e) number of text messages and emails; f) time spent using the smartphone; g) time spent on social media; and h) battery life.
Irritability | At entry (T0), 1-3 days after the last psychotherapeutic session (intervention group) OR 1-3 days after the last video is made available (active control group) (T1) and 30 days after these dates (T2)
  Changes in irritability reported by parents between T0 and T1, and T0 and T2, using the the Affective Reactivity Index (ARI), an index created to assess irritability, regarding their child. ARI is a 7 item scale (each scored with a 4 point likert scale), with higher scores corresponding to more severe irritability. It will be fulfilled by the blind assessor, in an interview with the main caregiver (through videoconference or phone call).
Parents satisfaction with the telepsychotherapeutic sessions | 1-3 days after the last psychotherapeutic session (intervention group only)
  Parents will be requested to fulfill an adapted version of the Telemedicine Satisfaction Questionnaire (intervention group only) to assess their satisfaction with this form of psychotherapy It will be fulfilled by the blind assessor, in an interview with the main caregiver (through videoconference or phone call).
primary measures of potential harm | At entry (T0), 1-3 days after the last psychotherapeutic session (intervention group) OR 1-3 days after the last video is made available (active control group) (T1) and 30 days after these dates (T2)
  emergence of suicidality in the child/adolescent reported by parents in T1 and T2, using 4 questions of the Mood and Feelings Questionnaire ("s/he thought that life wasn't worth living", "s/he thought about death or dying", "s/he thought his/her family would be better off without him/her", s/he thought about killing him/herself), regarding the past two weeks. It will be fulfilled by the blind assessor, in an interview with the main caregiver (through videoconference or phone call).
secondary measures of potential harm | At entry (T0), 1-3 days after the last psychotherapeutic session (intervention group) OR 1-3 days after the last video is made available (active control group) (T1) and 30 days after these dates (T2)
  worsening of the quality of family relationships.The family relationship subscale of the family impact module of the PedsQL will be completed by a caregiver at baseline and reassessed by the blind assessor in interviews (through videoconference or phone call) with the caregiver at T1 and T2.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme V Polanczyk, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto de Psiquiatria do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Background] American Academy of Child and Adolescent Psychiatry (AACAP) Committee on Telepsychiatry and AACAP Committee on Quality Issues. Clinical Update: Telepsychiatry With Children and Adolescents. J Am Acad Child Adolesc Psychiatry. 2017 Oct;56(10):875-893. doi: 10.1016/j.jaac.2017.07.008. Epub 2017 Jul 25. PMID 28942810
- [Background] DeSousa DA, Stringaris A, Leibenluft E, Koller SH, Manfro GG, Salum GA. Cross-cultural adaptation and preliminary psychometric properties of the Affective Reactivity Index in Brazilian Youth: implications for DSM-5 measured irritability. Trends Psychiatry Psychother. 2013;35(3):171-80. doi: 10.1590/s2237-60892013000300004. PMID 25923389
- [Background] Ebesutani C, Korathu-Larson P, Nakamura BJ, Higa-McMillan C, Chorpita B. The Revised Child Anxiety and Depression Scale 25-Parent Version: Scale Development and Validation in a School-Based and Clinical Sample. Assessment. 2017 Sep;24(6):712-728. doi: 10.1177/1073191115627012. Epub 2016 Feb 1. PMID 26834091
- [Background] Matcham F, Barattieri di San Pietro C, Bulgari V, de Girolamo G, Dobson R, Eriksson H, Folarin AA, Haro JM, Kerz M, Lamers F, Li Q, Manyakov NV, Mohr DC, Myin-Germeys I, Narayan V, Bwjh P, Ranjan Y, Rashid Z, Rintala A, Siddi S, Simblett SK, Wykes T, Hotopf M; RADAR-CNS consortium. Remote assessment of disease and relapse in major depressive disorder (RADAR-MDD): a multi-centre prospective cohort study protocol. BMC Psychiatry. 2019 Feb 18;19(1):72. doi: 10.1186/s12888-019-2049-z. PMID 30777041
- [Background] Oar EL, Johnco C, Ollendick TH. Cognitive Behavioral Therapy for Anxiety and Depression in Children and Adolescents. Psychiatr Clin North Am. 2017 Dec;40(4):661-674. doi: 10.1016/j.psc.2017.08.002. Epub 2017 Sep 19. PMID 29080592
- [Background] Varni JW, Sherman SA, Burwinkle TM, Dickinson PE, Dixon P. The PedsQL Family Impact Module: preliminary reliability and validity. Health Qual Life Outcomes. 2004 Sep 27;2:55. doi: 10.1186/1477-7525-2-55. PMID 15450120
- [Background] Woerner W, Fleitlich-Bilyk B, Martinussen R, Fletcher J, Cucchiaro G, Dalgalarrondo P, Lui M, Tannock R. The Strengths and Difficulties Questionnaire overseas: evaluations and applications of the SDQ beyond Europe. Eur Child Adolesc Psychiatry. 2004;13 Suppl 2:II47-54. doi: 10.1007/s00787-004-2008-0. PMID 15243786
- [Background] Yip MP, Chang AM, Chan J, MacKenzie AE. Development of the Telemedicine Satisfaction Questionnaire to evaluate patient satisfaction with telemedicine: a preliminary study. J Telemed Telecare. 2003;9(1):46-50. doi: 10.1258/135763303321159693. PMID 12641893
- [Derived] Casella CB, Farhat LC, Labbadia EM, Zuccolo PF, Fatori D, Argeu A, Salum GA, Polanczyk GV. Brief Internet-Delivered Cognitive-Behavioral Intervention for Children and Adolescents With Emotional Symptoms in Brazil: A Randomized Clinical Trial. J Adolesc Health. 2025 Sep;77(3):472-483. doi: 10.1016/j.jadohealth.2025.01.021. Epub 2025 Apr 2. PMID 40172510
- [Derived] Casella CB, Zuccolo PF, Sugaya L, de Souza AS, Otoch L, Alarcao F, Gurgel W, Fatori D, Polanczyk GV. Brief internet-delivered cognitive-behavioural intervention for children and adolescents with symptoms of anxiety and depression during the COVID-19 pandemic: a randomised controlled trial protocol. Trials. 2022 Oct 22;23(1):899. doi: 10.1186/s13063-022-06836-2. PMID 36273162